CLINICAL TRIAL: NCT03862456
Title: Clinical and Microbiological Comparison of Two Different Systemic Antimicrobials (Azithromycin Versus Metronidazole) as Adjuncts to Periodontal Surgery in the Treatment of P.Gingivalis Periodontitis Patients
Brief Title: Metronidazole vs Azithromycin in Periodontal Surgery for Patients Positive to Porphyromonas Gingivalis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATB1
Record Dates: First submitted 2019-02-20; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Periodontitis; Surgery
Keywords: Disease Progression; Microbiota; Periodontitis/surgery; Periodontitis/therapy; Periodontitis/drug effect; Periodontitis/drug therapy; Periodontal diseases/surgery; Periodontal diseases/therapy; Periodontal pocket/surgery; Periodontal pocket/therapy; Periodontal pocket/drug therapy; Azithromycin/therapeutic use; Metronidazole/therapeutic use; Azithromycin; Metronidazole; Porphyromonas gingivalis
MeSH Terms: conditions — Periodontitis; Disease Progression; Periodontal Diseases; Periodontal Pocket | interventions — Azithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subjects were randomly assigned to the treatment groups in ascending order according to a balanced distribution system through a computer generated random number design table (random block design). Randomization was balanced according to the smoking habit at the initial visit to ensure homogeneity in the treatment groups.
  The method of allocation concealment selected were opaque envelopes. The research coordinator was responsible for the randomization and allocation of patients.
  The 50 opaque envelopes (25 / group) were prepared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- azythromycin + periodontal surgery. (Experimental): Periodontal surgery + Azithromycin (500 mg every 24 h for 3 days).
  Interventions: Other: Azithromycin
- metronidazole + periodontal surgery (Active Comparator): Periodontal surgery + Metronidazole (500 mg every 8 h for 7 days).
  Interventions: Other: Metronidazole

INTERVENTIONS:
Other: Azithromycin — azithromycin (500 mg/24h/3 days)
  Arms: azythromycin + periodontal surgery.
Other: Metronidazole — metronidazole (500 mg/8h/7 days)
  Arms: metronidazole + periodontal surgery

SUMMARY:
The objective of this study is to determine whether, in patients with non treated periodontitis (stage III and IV) positive to Porphyromonas gingivalis, the use of systemic antimicrobials (metronidazole versus azithromycin) as an adjunctive treatment to periodontal surgery provides clinical and microbiological benefits.

DETAILED DESCRIPTION:
Design: randomized, parallel and triple blind clinical trial

Sample: Patients with periodontitis (stages III and IV) and positive to Porphyromonas gingivalis who potentially need periodontal surgery were recruited. 25 patients were randomized to the test group (periodontal surgery + azithromycin) and another 25 subjects to the control group (periodontal surgery + metronidazole).

Study visits:

* Examiner calibration
* Recruitment of patients. Screening. Data collection (clinical and microbiological variables).
* Phase I.

  * Non-surgical periodontal treatment (2 visits).
  * Reevaluation at 6 weeks. Data collection (clinical and microbiological variables). Identification of study candidate patients (Patients with probing pocket depth > 5 mm and positive to Porphyromonas gingivalis). Randomization of study groups.
* Phase II. Surgical periodontal treatment.

  * Periodontal surgery sessions. In the last surgery, the antibiotic test (azithromycin) or metronidazole (control) is administered according to randomization.
  * Suture removal 1 week after performing periodontal surgery. Data collection 1 week after antibiotic consumption with the last surgery (patient-centered variables on the side effects of antibiotics).
  * Re-evaluation of the surgical phase at 6 weeks after the last surgery session. Data collection (clinical variables).
* Phase III. Periodontal maintenance.

  * Maintenance 1 (3 months post surgery). Data collection (Clinical and microbiological variables).
  * Maintenance 2 (6 months post surgery). Data collection (Clinical and microbiological variables).
  * Maintenance 3 (9 months post surgery). Data collection (Clinical variables).
  * Maintenance 4 (12 months post surgery). Data collection (Clinical and microbiological variables).
  * Maintenance 5 (4 years post surgery). Data collection (Clinical and microbiological variables).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of periodontitis (stages III or IV) that may require periodontal surgery
* Have at least 10 teeth in function, excluding third molars.
* Present locations with probing depth (PS)> 6 mm in at least 30% of the teeth.
* Present radiographic evidence of moderate-severe bone loss in at least 30% of the dentition.
* Detection of P. gingivalis in subgingival samples taken at the screening visit as well as in the post-scaling and root planning visit and processed by culture.
* Systemically healthy patients.

Exclusion Criteria:

* Pregnant or lactating women.
* Presenting systemic pathology and / or taking medication that may affect the periodontal situation and / or patients requiring antibiotic prophylaxis.
* Have received systemic antimicrobial treatment in the previous 6 months.
* Have received periodontal treatment in the 6 months prior to the beginning of the study.
* Patients allergic to metronidazole, or to any of the components of commercial formulations thereof (Flagyl®).
* Patients allergic to azithromycin, or to any of the components of commercial formulations thereof (Zithromax®).
* Patients who refuse to sign the informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth (PPD) | At 6 weeks after periodontal surgery
  Full mouth measurement at 6 sites per tooth, with a manual periodontal probe University North Carolina 15 (UNC-15 mm)

SECONDARY OUTCOMES:
Probing pocket depth (PPD) | At the beginning of the study, 6 weeks after scaling and root planning (Reevaluation phase I), 6 weeks after the last surgery session (Reevaluation Phase II) and during the maintenance Phase III (3, 6, 9, 12 and 48 months after periodontal surgery)
  Full mouth measurement at 6 sites per tooth, with a manual periodontal probe UNC-15 mm
Gingival Recession (REC) | At the beginning of the study, 6 weeks after scaling and root planning (Reevaluation phase I), 6 weeks after the last surgery session (Reevaluation Phase II) and during the maintenance Phase III (3, 6, 9, 12 and 48 months after periodontal surgery)
  Full mouth measurement at 6 sites per tooth, with a manual periodontal probe UNC-15 mm
Plaque index (PlI) | At the beginning of the study, 6 weeks after scaling and root planning (Reevaluation phase I), 6 weeks after the last surgery session (Reevaluation Phase II) and during the maintenance Phase III (3, 6, 9, 12 and 48 months after periodontal surgery)
  Full mouth measurement at 6 sites per tooth, with a manual periodontal probe UNC-15 mm
Gingival index (GI) | At the beginning of the study, 6 weeks after scaling and root planning (Reevaluation phase I), 6 weeks after the last surgery session (Reevaluation Phase II) and during the maintenance Phase III (3, 6, 9, 12 and 48 months after periodontal surgery)
  Full mouth measurement of the bleeding on probing at 6 sites per tooth, with a manual periodontal probe UNC-15 mm
Furcations | At the beginning of the study, 6 weeks after scaling and root planning (Reevaluation phase I), 6 weeks after the last surgery session (Reevaluation Phase II) and during the maintenance Phase III (3, 6, 9, 12 and 48 months after periodontal surgery)
  Measurement of furcations with a manual periodontal probe UNC-15 mm
Clinical attachment level (CAL) | At the beginning of the study, 6 weeks after scaling and root planning (Reevaluation phase I), 6 weeks after the last surgery session (Reevaluation Phase II) and during the maintenance Phase III (3, 6, 9, 12 and 48 months after periodontal surgery)
  Full mouth measurement at 6 sites per tooth, with a manual periodontal probe UNC-15 mm
Total bacterial counts | At the beginning of the study, 6 weeks after scaling and root planning (Reevaluation phase I) and during the maintenance Phase III (3, 6, 12 and 48 months after periodontal surgery)
  A microbiological sample is taken with sterilized paper points from the gingival crevicular fluid and the total bacterial counts (expressed in total colony-forming units) are analyzed by culture.
Percentage of periodontal pathogens | At the beginning of the study, 6 weeks after scaling and root planning (Reevaluation phase I) and during the maintenance Phase III (3, 6, 12 and 48 months after periodontal surgery)
  Determination of the percentage of the following periodontal pathogens:
  * Porphyromonas gingivalis
  * Tannerella forsythia
  * Aggregatibacter actinomycetemcomitans
  * Prevotella intermedia
  * Fusobacterium nucleatum
  * Eikenella corrodens
  * Campylobacter rectus
  * Capnocytophaga sp.
  * Enterobacter sp.
Counts of periodontal pathogens | At the beginning of the study, 6 weeks after scaling and root planning (Reevaluation phase I) and during the maintenance Phase III (3, 6, 12 and 48 months after periodontal surgery)
  Determination of the following periodontal pathogens: Porphyromonas gingivalis
  * Tannerella forsythia
  * Aggregatibacter actinomycetemcomitans
  * Prevotella intermedia
  * Fusobacterium nucleatum
  * Eikenella corrodens
  * Campylobacter rectus
  * Capnocytophaga sp.
  * Enterobacter sp.
Appearance of side effects after taking antibiotic | 1 week after antibiotic consumption
  The patient was asked if he had side effects after taking antibiotic (Yes / No)
Type of adverse effect after taking antibiotic | 1 week after antibiotic consumption
  The patient was asked to write freely on a form the type of side effect suffered
Degree of affectation | 1 week after antibiotic consumption
  The patient was asked to categorize the degree of affectation (mild, moderate or severe) of the secondary effect of the antibiotic if it had appeared.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, Study Director — University Complutense Madrid (UCM)
Locations (1):
- Faculty of Dentistry, Univesity Complutense, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No